CLINICAL TRIAL: NCT03201536
Title: ZipLine Incision Approzimation Vs. Suture:Zips3 Physician Preference Study
Brief Title: ZipLine Incision Approximation Verses Suture:ZIPS3 Physician Preference Study
Acronym: ZIPS3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-002-12
Record Dates: First submitted 2012-05-21; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Wounds and Injuries
Keywords: ZipLine3 device vs. conventional sutures
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sutures (Active Comparator): zipLine3 device verses conventional sutures
  Interventions: Device: conventional Suture
- Zip3 Device (Active Comparator)
  Interventions: Device: Zip3

INTERVENTIONS:
Device: conventional Suture — Sutures
  Other Names: stitches,PeriStrips
  Arms: sutures
Device: Zip3 — wound closure device
  Arms: Zip3 Device

SUMMARY:
Zipline incision approximation vs. Suture -- zips 3 study. A prospective, multi-site, non-blinded, randomized controlled, study designed to evaluate user preferences associated with use of the zipline 3 system versus conventional suturing for incision closure.

DETAILED DESCRIPTION:
The objective of this study is to evaluate user preferences associated with the ZipLine 3 system versus conventional suture placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 75 years of age

   * In generally good health
   * Willing to be evaluated in 5-14 days and 3-months post op
2. Patient requiring a non-emergent skin incision or biopsy

   * Maximum excision size 1.5x3.0 cm
   * Requiring 4-0 or smaller suture for closure
   * In area of body trunk or extremities with low mobility and tension

Exclusion Criteria:

1. Facial Incisions or incisions in high stress or tension areas
2. Previously diagnosed peripheral vascular disease
3. Insulin-dependent diabetes mellitus
4. Known bleeding diathesis
5. Known personal or family history of keloid formation or scar hypertrophy
6. Known allergy or hypersensitivity to adhesives
7. Presently taking steroids, immune stimulants, beta blockers, or anticoagulants
8. Atrophic skin deemed clinically prone to blistering
9. Any skin disorder affecting wound healing
10. Incisions requiring dermal sutures
11. Any other condition that in the opinion of the investigator would make a particular patient unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Wound healing | 3-month
  Wound healing as judged by the CVAS (Cosmetic Visual Analogue Scale) wound healing scale

SECONDARY OUTCOMES:
time of procedure | immediately
  Time it takes to use device

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Parret, MD, Principal Investigator — Plastic Surgery Institute of Northern California; Landon Clark, MD,MPH, Principal Investigator — Palo Alto Medical Foundation; Stanley P Leong, MD,FACS, Principal Investigator — California Pacific Medical Center
Locations (3):
- United States (3):
  - Palo Alto Medical Foundation, Palo Alto, California
  - Plastic Surgery Institute of Northern California, San Francisco, California
  - California Pacific Medical Center, San Francisco, California